CLINICAL TRIAL: NCT03838497
Title: Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine Among HIV-infected Adults in the Era of Highly Active Antiretroviral Therapy: Analysis Stratified by CD4 T-cell Count
Brief Title: Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine Among HIV-infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Joon Young Song, Professor, Korea University Guro Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014GR0014
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Streptococcal Pneumonia; HIV/AIDS
MeSH Terms: conditions — Pneumonia; Acquired Immunodeficiency Syndrome | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HIV-infected subjects with CD4 T-cell counts <350 cells/µL (Active Comparator): Intervention to be administered: Prevenar13
  Interventions: Biological: Prevenar13
- HIV-infected subjects with CD4 T-cell counts ≥350 cells/µL (Active Comparator): Intervention to be administered: Prevenar13
  Interventions: Biological: Prevenar13

INTERVENTIONS:
Biological: Prevenar13 — Prevenar13 for both arms

SUMMARY:
HIV-infected patients are 30- to 100-fold more susceptible to invasive pneumococcal diseases. Pneumococcal vaccination is the best way to decrease the large pneumococcal disease burden, but the optimal timing of vaccination is still unclear. HIV-infected subjects aged ≥ 18 years were recruited and divided into two age-matched groups: group 1 (subjects with CD4 T-cell counts ≥350 cells/µL) and group 2 (subjects with CD4 T-cell counts <350 cells/µL). Multiplex opsonophagocytic killing assay was used to compare immunogenicity after the immunization of 13-valent pneumococcal conjugate vaccine (PCV13).

DETAILED DESCRIPTION:
This single-center, open-label non-randomized clinical trial was conducted at Korea University Guro Hospital from April 2015 to January 2017. Based on the CD4 T-cell counts at the time of study enrollment, HIV-infected subjects aged ≥ 18 years were divided into two groups, group 1 (subjects with CD4 T-cell counts ≥350 cells/µL) and group 2 (subjects with CD4 T-cell counts <350 cells/µL).

The primary objective of the study was to demonstrate that the immune responses to PCV13 serotypes in Group 2 (CD4 T-cell counts <350 cells/µL) were not inferior to those in Group 1 (CD4 T-cell counts ≥350 cells/µL) at one month after vaccination. In addition, the safety profiles of PCV13 were compared between two study groups.

HIV-infected subjects aged ≥ 18 years with stable underlying diseases (≥ 4 weeks on HAART) were eligible for this study. All available subjects with low CD4 T-cell counts (<350 cells/µL, group 2) were recruited, and age/visit day-matched controls with high CD4 T-cell counts (≥350 cells/µL, group 1) were enrolled. The exclusion criteria were as follows: 1) a history of pneumococcal infection within the recent five years, 2) previous pneumococcal vaccination, 3) current opportunistic infections, 4) known immunodeficiency other than HIV infection and 5) coagulation disorders.

The study was approved by the ethics committee of Korea University Guro Hospital (IRB No. 2014GR0014) and was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice. Informed consent was taken for all participants before enrollment. Venous blood samples of 10 mL were collected on day 0 and post-vaccination day 28 ± 7.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infeted subjects who received antiretroviral therapy for ≥ 4 weeks

Exclusion Criteria:

* a history of pneumococcal infection within the recent five years
* previous pneumococcal vaccination
* current opportunistic infections
* known immunodeficiency other than HIV infection
* coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Opsonophagocytic assay (OPA) titers for PCV13 | Outcome measure will be assessed at two points (baseline and 28 ± 7 days after vaccination).
  OPA geometric mean titers for 13 PCV13 serotypes with corresponding 2-sided 95% confidence intervals between groups receiving PCV 13 and then compare the results

SECONDARY OUTCOMES:
Frequency and duration of local and systemic adverse events | All participants will be followed until 4 weeks after vaccination
  The safety profiles of co-administration of Fluad and PCV13 will be compared to those of single vaccination.

IPD SHARING:
Plan to Share IPD: No